CLINICAL TRIAL: NCT06934993
Title: Comparison of Bidirectional Palpation Test and Transit Time Flow Measurement for LIMA-LAD Graft Patency
Status: Completed | Type: Observational
Sponsor: Abdulgani Orhun YENİGÜN (Other)
Responsible Party: Sponsor-Investigator, Abdulgani Orhun YENİGÜN, Principal Investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Other Study IDs: E-83045809-604.01-1014609
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Coronary Arterial Disease (CAD); Coronary Artery Bypass; LIMA; Graft Patency; LAD (Left Anterior Descending) Coronary Artery Stenosis; Saphenous Vein Graft Patency; LIMA-LAD ANASTOMOSIS; LIMA GREFT PATENCY
Keywords: GRAFT PATENCY; LIMA-LAD ANATOMOSIS; LIMA GRAFT PATENCY; SAPHENOUS VEİN GRAFT PATENCY; CABG
MeSH Terms: conditions — Leukocyte adhesion deficiency type 1; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elective CABG Patients with LIMA-to-LAD Grafts: This cohort consists of patients who underwent elective coronary artery bypass grafting (CABG) with a left internal mammary artery (LIMA) to left anterior descending artery (LAD) anastomosis, and who were evaluated using intraoperative TTFM and BDPT, followed by early postoperative CTA imaging.

SUMMARY:
The most important factor determining mortality and morbidity after coronary artery bypass graft (CABG) surgery is graft patency. The LIMA-LAD anastomosis is the most crucial anastomosis because it's revascularizing the most important and large region of the heart, has superior long-term graft patency rates and is considered the gold standard for CABG. Therefore, ensuring the patency of the LIMA-LAD anastomosis is vital for both early and late outcomes. The bidirectional palpation test (BPT), developed in our clinic to assess graft patency, is a subjective test, yet it is simple and reliable. Additionally, transit time flow meter (TTFM) measurements have also been performed. In this study, the efficacy of BPT and the results of TTFM measurements were compared by examining graft patency through early-period coronary CT angiography (CCTA).

DETAILED DESCRIPTION:
STUDY DESIGN This study was designed as a retrospective-prospective hybrid cohort study. The study population was selected among patients who underwent LIMA-LAD anastomosis during CABG surgery at our clinic. Patients who wished to participate in the study gave informed consent by signing a preoperative consent form. Intraoperative BPT (Bidirectional Palpation Test) results and TTFM (Transit-Time Flow Measurement) values were recorded and compared with the early postoperative period (first month) CTCA (Coronary Tomography Angiography) findings. Data from 23 of the 73 patients included in the study were obtained retrospectively, while data from the remaining 50 patients were collected prospectively. All procedures performed on patients throughout the study were conducted in accordance with ethical standards, and patient information was kept confidential.

ETHICS COMMITTEE This study was conducted in accordance with the guidelines of the Clinical Research Ethics Committee of Istanbul University Cerrahpaşa and the principles outlined in the Declaration of Helsinki. In this retrospective-prospective hybrid cohort study, all data were anonymized. Throughout the study process, participant privacy and the protection of personal data were prioritized. Patient confidentiality was ensured in full compliance with ethical standards and relevant legal regulations. This approach ensured that ethical principles were maintained throughout the research process and that participants' rights were protected.

PATIENT SELECTION A total of 73 patients who underwent elective isolated CABG surgery or CABG in combination with other procedures such as valve surgery or ascending aorta surgery and gave informed consent were included in the study. However, 43 patients were excluded for reasons such as refusing to participate postoperatively, death in the early postoperative period (3 patients), or conditions like elevated postoperative creatinine that precluded CTCA. As a result, 73 patients remained in the final analysis, and a total of 73 LIMA grafts were evaluated. To minimize the impact of the anastomosis technique and quality on the study outcomes, all surgeries were performed by the same surgical team.

INTRAOPERATIVE PLANNING Following standard surgical preparation under general anesthesia, patients were properly draped. After a median sternotomy, pedicled LIMA and saphenous vein grafts were harvested. The patient was heparinized, and the Activated Clotting Time (ACT) was raised above 450 seconds. After opening the pericardium, arterial cannulation of the aorta and venous cannulation of the right atrium were performed, and cardiopulmonary bypass (CPB) was initiated. Diastolic arrest was achieved using antegrade cold Del Nido cardioplegia after applying the aortic cross-clamp. Once the distal anastomoses were completed, the cross-clamp was removed. Proximal anastomoses were performed on the beating heart using a side clamp. After de-airing and gradual reduction of flow, CPB was discontinued. Once the heart resumed circulation, a segment of the LIMA was stripped of surrounding tissue for measurement. With mean arterial pressure maintained above 60 mmHg, TTFM and ÇYPT assessments of the LIMA-LAD anastomosis were performed. If the BPT result on LIMA was positive and the flow rate and PI measured by TTFM were within acceptable ranges, TTFM measurements of the saphenous vein grafts were then conducted. Once acceptable TTFM values were confirmed for the SVGs as well, hemodynamic and arrhythmia monitoring continued. If hemodynamics remained stable, protamine was administered to neutralize heparin, and the heart was decannulated. After ensuring hemostasis, mediastinal and left thoracic drains were placed. Temporary epicardial pacing wires were inserted, the sternum was closed with wire sutures, and the subcutaneous and skin layers were closed anatomically to complete the surgery.

BIDIRECTIONAL PALPATION TEST AND TTFM MEASUREMENTS In this method, after completing the anastomoses, CPB is temporarily discontinued to create a pulse pressure, and a segment on the LIMA with a palpable pulse is identified. In the first step, the distal part of the palpated segment is occluded using a bulldog clamp or the surgeon's hand, and if the pulse persists, proximal flow is confirmed. This assesses the antegrade flow from the subclavian artery into the LIMA. In the second step, the distal occlusion is released, and a bulldog clamp or manual occlusion is applied proximally to the palpated area. If the pulse remains palpable, retrograde flow and indirectly, the patency of the LIMA-LAD anastomosis are confirmed . Due to venous valve structures preventing backflow, BPT cannot routinely be used on SVGs. However, in cases of valve insufficiency causing regurgitation in the graft, SVGs can also be evaluated using BPT.

DATA RECORDING Data collection was carried out in three stages. In the first stage, preoperative data were obtained by reviewing patient files. In the second stage, intraoperative Bidirectional Palpation Test results and TTFM (Transit-Time Flow Measurement) values were evaluated and recorded by the surgeon. During postoperative follow-ups, patients were called in for a check-up in the first week after discharge, and blood tests-including renal function tests-were performed. Based on the test results, patients deemed suitable for CTCA (Coronary Tomography Angiography) were scheduled for imaging within the first postoperative month, and their imaging procedures were monitored. In the third stage, CTCA results were reported by radiologist and recorded. Grafts showing more than 50% luminal stenosis were considered occluded. These steps were designed to enhance the accuracy and reliability of the data.

PATIENT FOLLOW-UP Patients included in the study were closely monitored in the cardiovascular surgery intensive care unit and on the ward during the postoperative period. Upon discharge, patients were prescribed necessary medications and provided with relevant recommendations. To prevent graft occlusion, all patients were routinely prescribed either dual or single antiplatelet therapy, cholesterol-lowering agents, beta-blockers to prevent arrhythmias, and anticoagulants when necessary. Compliance with these treatments was closely monitored. Each medication's purpose, possible side effects, and interactions with other drugs were explained to the patients in detail. As part of secondary prevention, risk factors such as obesity, smoking, hyperlipidemia, diabetes, and hypertension were addressed through both pharmacological treatment and lifestyle modifications. Routine follow-ups were scheduled on postoperative day 7, and at 1, 6, and 12 months using laboratory tests and imaging techniques.

STATISTICAL ANALYSIS The study data were analyzed using the SPSS 25.0 statistical software package. For descriptive analyses, frequency distributions and percentages were calculated, means were presented with standard deviations, and medians were shown with minimum and maximum values. Since the data did not follow a normal distribution, the Mann-Whitney U test and Kruskal-Wallis test were used for comparisons between groups. The relationships between categorical variables were evaluated using the Pearson Chi-square test. In 2x2 tables, when the expected value in at least one cell was less than 5, Fisher's exact Chi-square test was applied, and when any observed value ranged between 5 and 20, the Yates-corrected Chi-square test was used. ROC analysis was performed to determine cut-off values for certain variables. A p-value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Elective Isolated CABG Surgery: Patients undergoing elective isolated coronary artery bypass grafting (CABG).
2. CABG with Additional Cardiac Surgery: Patients who had CABG surgery in conjunction with other cardiac procedures.
3. Informed Consent: Patients who provided informed consent to participate in the study.
4. Postoperative Follow-Up: Patients who were followed up postoperatively and completed the necessary evaluations.
5. CABG patients whose renal functions are suitable for CTA

Exclusion Criteria:

Refusal to Participate: Patients who did not wish to participate in the study after being approached.

Death in Early Postoperative Period: Patients who died in the early postoperative period (3 patients).

Inability to Perform CABG: Patients for whom CABG could not be performed due to postoperative complications (e.g., elevated creatinine levels leading to inability to perform CABG, 43 patients).

Patients in whom CT angiography is not appropriate: Such as acute or chronic renal failure

Ages: 41 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 73 patients who underwent coronary artery bypass surgery (CABG) and LIMA-LAD anastomosis
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdulgani Orhun yenigün, Principal Investigator — İstanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine
Locations (1):
- İstanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning after the publication of results and ending a year later.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent rewiev committee identified for this purpose
URL: https://docs.google.com/document/u/0/

REFERENCES:
- See also: Related Info — https://docs.google.com/document/d/18BaS1fHrkVkHIiYzNlN0CmgH7mLS9MH2H82qL_TXMsA/edit?tab=t.0
- Available data/document: Study Protocol — https://docs.google.com/document/d/18BaS1fHrkVkHIiYzNlN0CmgH7mLS9MH2H82qL_TXMsA/edit?tab=t.0 — The data will be uploaded three months after the publication of the study. The data is not currently available at the provided address.
- Available data/document: Individual Participant Data Set — https://docs.google.com/spreadsheets/d/1wNK5vDSm42LuTVoIUTiuYG_Yg_b2tGHBi1PKytJVMNw/edit?usp=sharing — The data will be uploaded three months after the publication of the study. The data is not currently available at the provided address.
- Available data/document: Informed Consent Form — https://docs.google.com/document/d/1F8ermx5WFwjpxtn4MubaZDkew90csOJMbjbKOXvCgC0/edit?usp=sharing — The data will be uploaded three months after the publication of the study. The data is not currently available at the provided address.
- Available data/document: Statistical Analysis Plan — https://docs.google.com/document/d/1nG06s9_mVy9alLULhhv0LBmW4YkqVBX1RBXj8GoaGXQ/edit?usp=sharing — The data will be uploaded three months after the publication of the study. The data is not currently available at the provided address.
- Available data/document: Clinical Study Report — https://docs.google.com/document/d/17UWmXMrss0xVXFFsI-ulf6aGNU3tHCWMr34yhpWYiNA/edit?usp=sharing — The data will be uploaded three months after the publication of the study. The data is not currently available at the provided address.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 116 patients who underwent elective isolated CABG surgery or CABG in combination with other procedures such as valve surgery or ascending aorta surgery and gave informed consent were included in the study. The first patient was enrolled in the study on August 31, 2023 while the last patient was enrolled on August 27, 2024.
Pre-assignment Details: Patients were excluded for reasons such as refusing to participate postoperatively, death in the early postoperative period , or conditions like elevated postoperative creatinine that precluded CTCA.
Period: Overall Study
Arm/Group | Elective CABG Patients With LIMA-to-LAD Grafts
Started | 116
Completed | 73
Not Completed | 43
Not completed — Withdrawal by Subject | 29
Not completed — elevated postoperative creatinine level | 11
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Elective CABG Patients With LIMA-to-LAD Grafts
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.25 (7.76)
Age, Continuous [Median (Full Range); unit: years] | 58 [41 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 73
Diabetes Mellitus (DM) [Count of Participants; unit: Participants] | 40
Peripheral Artery Disease (PAD) [Count of Participants; unit: Participants] | 6
Smoking [Count of Participants; unit: Participants] | 50
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 28.11 (3.44)
Hypertension [Count of Participants; unit: Participants] | 53
Body Mass Index (BMI) [Median (Full Range); unit: kg/m²] | 27.72 [21.48 to 40.82]

OUTCOME MEASURES:

1. Primary Outcome: Reliability of Bidirectional Palpation Test (BPT) in Evaluating LIMA-LAD Graft Patency
Description: The reliability of the Bilateral Palpation Test (BPT) in evaluating LIMA-LAD graft patency was assessed. As detailed in the Study Description section, participants were evaluated intraoperatively as BPT-positive or BPT-negative. Grafts were considered patent in BPT-positive participants and occluded in those with negative findings. In the early postoperative period, contrast-enhanced coronary CT angiography (CCTA), a validated method for assessing graft patency, was performed. The correlation between CCTA and BPT results was then analyzed to evaluate the reliability of the BPT.
Time Frame: Postoperative first month.
Population: The number of patients with graft occlusion among 73 patients who participated in the study was examined. Then, BPT negativity in patients with graft occlusion and BPT positivity in patients with patent grafts were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Elective CABG Patients With LIMA-to-LAD Grafts
Number analyzed (Participants) | 73
Participants
  Patients with LIMA-LAD graft occlusion (CCTA) | 2
  Patients with negative BPT | 2
  Patients with BPT negativity and LIMA-LAD graft occlusion (CCTA) | 2
  BPT negativity in patients with LIMA-LAD graft occlusion (CCTA): number analyzed (Participants) | 2
  BPT negativity in patients with LIMA-LAD graft occlusion (CCTA) | 2
  BPT positivity in patients with patent LIMA-LAD grafts (CCTA): number analyzed (Participants) | 71
  BPT positivity in patients with patent LIMA-LAD grafts (CCTA) | 71
Statistical Analysis 1: Comparison: Elective CABG Patients With LIMA-to-LAD Grafts; In LIMA-LAD cases, when the post hoc power analysis results for the relationship between graft patency and flow rate were examined, the effect size was found to be 0.836, with an alpha error level set at 0.05. The statistical power of the study was determined to be 99.99%; Test type: Superiority; p < 0.001, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05

2. Primary Outcome: Reliability of TTFM in Evaluating LIMA-LAD Graft Patency
Description: Mean Graft Flow (MGF) and Pulsatility Index (PI) were used in this study as TTFM parameters for evaluating graft patency. In the literature, there is no clear consensus on cut-off values for these parameters. Therefore, the values commonly used in the literature were statistically analyzed, and the values that gave the most significant results with our data were accepted as cut-off values. These cut-off values were determined to be 10 ml/min for MGF and 4.5 for PI.
Time Frame: Postoperative first month
Population: While evaluating graft patency in the 73 patients included in the study, the correlation of MGF <10 ml/min and PI >4.5 measurements was analyzed both individually and in combination among patients with graft occlusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Elective CABG Patients With LIMA-to-LAD Grafts
Number analyzed (Participants) | 73
Participants
  Patients with LIMA-LAD graft occlusion | 2
  Patients with measured MGF<10ml/min | 3
  Patients with measured PI>4,5 | 23
  Patients with measured MGF<10ml/min and PI>4,5 | 3
  Patients with measured MGF<10ml/min and PI<4,5 or MGF>10 and PI>4,5 | 20
  Patients with measured MGF<10ml/min with LIMA-LAD graft occlusion: number analyzed (Participants) | 2
  Patients with measured MGF<10ml/min with LIMA-LAD graft occlusion | 2
  Patients with measured MGF>10ml/min with patent LIMA-LAD graft: number analyzed (Participants) | 71
  Patients with measured MGF>10ml/min with patent LIMA-LAD graft | 70
  Patients with measured PI>4,5 with LIMA-LAD graft occlusion: number analyzed (Participants) | 2
  Patients with measured PI>4,5 with LIMA-LAD graft occlusion | 2
  Patients with measured PI<4,5 with patent LIMA-LAD graft: number analyzed (Participants) | 71
  Patients with measured PI<4,5 with patent LIMA-LAD graft | 50
  Patients with measured MGF<10ml/min and PI>4,5 with LIMA-LAD graft occlusion: number analyzed (Participants) | 2
  Patients with measured MGF<10ml/min and PI>4,5 with LIMA-LAD graft occlusion | 2
Statistical Analysis 1: Comparison: Elective CABG Patients With LIMA-to-LAD Grafts; In all cases, when the post hoc power analysis results for the relationship between graft patency and flow rate were examined, the effect size was found to be 0.836, with an alpha error level set at 0.05. The statistical power of the study was determined to be 99.99%; Test type: Superiority; p = 0.001, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05
Statistical Analysis 2: Comparison: Elective CABG Patients With LIMA-to-LAD Grafts; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.096, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05
Statistical Analysis 3: Comparison: Elective CABG Patients With LIMA-to-LAD Grafts; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05

3. Secondary Outcome: Correlation Between Intraoperative TTFM and BPT Results
Description: Mean Graft Flow (MGF) and Pulsatility Index (PI) were used in this study as TTFM parameters for evaluating graft patency. In the literature, there is no clear consensus on cut-off values for these parameters. Therefore, the values commonly used in the literature were statistically analyzed, and the values that gave the most significant results with our data were accepted as cut-off values. These cut-off values were determined to be 10 ml/min for MGF and 4.5 for PI. LIMA-LAD graft patency was considered compromised when MGF was <10 ml/min and/or PI was >4.5, whereas an MGF >10 ml/min and/or PI <4.5 was interpreted in favor of graft patency.
Time Frame: postoperative first month.
Population: This outcome was assessed only in a subgroup of 2 patients who had negative BPT. Therefore, the number of participants analyzed is lower than the total study population (N=73).
Measure: Count of Participants; unit: Participants
Groups:
- TTFM Parameters in Patients With Negative BPT: This cohort consists of patients who underwent elective coronary artery bypass grafting (CABG) with a left internal mammary artery (LIMA) to left anterior descending artery (LAD) anastomosis, and who were evaluated using intraoperative TTFM and BDPT, followed by early postoperative CTA imaging.
Arm/Group | TTFM Parameters in Patients With Negative BPT
Number analyzed (Participants) | 2
Participants
  The rate of MGF <10 mL/min among patients with a negative BPT. | 2
  The rate of PI>4.5 among patients with a negative BPT. | 2
Statistical Analysis 1: Comparison: TTFM Parameters in Patients With Negative BPT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05
Statistical Analysis 2: Comparison: TTFM Parameters in Patients With Negative BPT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.096, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05

4. Secondary Outcome: The Correlation of SYNTAX 1 and SYNTAX 2 Risk Scores With LIMA-LAD Graft Patency Was Evaluated.
Description: The correlation between preoperatively calculated SYNTAX 1 and SYNTAX 2 risk scores and LIMA-LAD graft patency, TTFM measurements and BPT was demonstrated. The SYNTAX I and SYNTAX II scores are risk assessment tools used to guide treatment decisions in patients with complex coronary artery disease. The SYNTAX I score is based solely on the anatomical complexity of coronary lesions observed during angiography. It categorizes patients into three risk groups: low (0-22), intermediate (23-32), and high (≥33).Higher SYNTAX I scores are associated with more complex coronary artery disease and worse clinical outcomes, often favoring coronary artery bypass grafting (CABG) over percutaneous coronary intervention (PCI). The SYNTAX II score combines anatomical factors with clinical variables such as age, gender, left ventricular ejection fraction, creatinine clearance, and the presence of comorbidities like COPD and peripheral artery disease. This comprehensive score provides a personalized risk
Time Frame: postoperative first month.
Population: The distributions of SYNTAX I and II scores were analyzed in patients with occluded grafts, MGF <10 ml/min and negative BPT.
Measure: Count of Participants; unit: Participants
Arm/Group | Elective CABG Patients With LIMA-to-LAD Grafts
Number analyzed (Participants) | 73
Participants
  SYNTAX I score: Low score | 18
  SYNTAX I score: Interm score | 29
  SYNTAX I score: High score | 26
  SYNTAX II score: Low score | 33
  SYNTAX II score: Interm score | 28
  SYNTAX II score: High score | 12
  SYNTAX I score distribution in patients with occluded LIMA-LAD grafts: number analyzed (Participants) | 2
  SYNTAX I score distribution in patients with occluded LIMA-LAD grafts: Low score | 2
  SYNTAX I score distribution in patients with occluded LIMA-LAD grafts: Interm score | 0
  SYNTAX I score distribution in patients with occluded LIMA-LAD grafts: High score | 0
  SYNTAX II score distribution in patients with occluded LIMA-LAD grafts: number analyzed (Participants) | 2
  SYNTAX II score distribution in patients with occluded LIMA-LAD grafts: Low score | 1
  SYNTAX II score distribution in patients with occluded LIMA-LAD grafts: Interm score | 1
  SYNTAX II score distribution in patients with occluded LIMA-LAD grafts: High score | 0
  SYNTAX I score distribution in patients with MGF<10 ml/min: number analyzed (Participants) | 3
  SYNTAX I score distribution in patients with MGF<10 ml/min: Low score | 3
  SYNTAX I score distribution in patients with MGF<10 ml/min: Interm score | 0
  SYNTAX I score distribution in patients with MGF<10 ml/min: High score | 0
  SYNTAX I score distribution in patients with BPT negativity: number analyzed (Participants) | 2
  SYNTAX I score distribution in patients with BPT negativity: Low score | 2
  SYNTAX I score distribution in patients with BPT negativity: Interm score | 0
  SYNTAX I score distribution in patients with BPT negativity: High score | 0
Statistical Analysis 1: Comparison: Elective CABG Patients With LIMA-to-LAD Grafts; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.04, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05
Statistical Analysis 2: Comparison: Elective CABG Patients With LIMA-to-LAD Grafts; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.679, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05
Statistical Analysis 3: Comparison: Elective CABG Patients With LIMA-to-LAD Grafts; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.011, Chi-squared — Statistical significance was defined as cases where the p-value was below 0.05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 months postoperatively.
Description: Adverse events were monitored in all 116 participants who underwent CABG surgery and were enrolled in the study. No serious or non-serious adverse events were observed during the postoperative period. However, 3 early postoperative deaths occurred before CT angiography could be performed. These were reported under all-cause mortality
Arm/Group | Elective CABG Patients With LIMA-to-LAD Grafts
All-Cause Mortality (participants affected / at risk) | 3/116
Serious Adverse Events (participants affected / at risk) | 0/116
Other Adverse Events (participants affected / at risk) | 11/116
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elective CABG Patients With LIMA-to-LAD Grafts (N=116)
Renal dysfunction (Renal and urinary disorders) | 11 (11) — Mild to moderate elevations in creatinine were observed in 11 participants, leading to exclusion from postoperative CT imaging. These events were transient, did not require hospitalization or dialysis.

LIMITATIONS AND CAVEATS:
The number of patients participating in the study was limited because the study was single-center and its duration was determined as 1 year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT06934993/Prot_000.pdf
  • Informed Consent Form (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT06934993/ICF_001.pdf